CLINICAL TRIAL: NCT05437497
Title: Safety and Efficacy Evaluation of Remimazolam for Endoscopic Ultrasound-guided Fine Needle Aspiration/Biopsy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Third Xiangya Hospital of Central South University (Other)
Responsible Party: Principal Investigator, wang xiaoyan, Doctor, The Third Xiangya Hospital of Central South University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: EUS-FNA-2022-01
Record Dates: First submitted 2022-06-23; First posted 2022-06-29 (Actual); Last update posted 2022-06-29 (Actual); Status verified 2022-06

CONDITIONS: Endoscopic Ultrasonography-guided Fine Needle Aspiration; Sedation Complication; Remimazolam
Keywords: Endoscopic ultrasound-guided fine needle aspiration; Sedation Complication; remimazolam
MeSH Terms: interventions — remimazolam; Propofol

STUDY DESIGN:
Intervention Model Description: The experimental group was sedated with remimazolam, and the control group was sedated with propofol;
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Care provider(anesthesiologist) cannot be blinded for different appearance of propofol and remimazolam.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Remimazolam group (Experimental): 1. Background oxycodone injection: Slowly inject oxycodone(0.05mg/kg) intravenously. Three minutes (± 1min) after the end of oxycodone injection , begin sedation induction as follows.
  2. Sedation induction before EUS-FNA/FNB: the initial dose of remimazolam is 0.15-0.2 mg/kg, and the intravenous injection time is about 1 minute. If the subject's MOAA/S score is 1 point or below after the initial dose, EUS-FNA/FNB can be started; if the degree of sedation is insufficient, additional remimazolam(0.05 mg/kg each time) is allowed. The injection time of additional remimazolam is not less than 15 seconds, and the time interval between each additional administration is ≥ 2 minutes.
  3. Maintenance of sedation: In order to maintain the MOAA/S≤1, the investigator can decide to add remimazolam 0.05mg/kg each time, and the intravenous injection time should not be less than 15 seconds, with an additional administration interval of ≥ 2 minutes.
  Interventions: Drug: Remimazolam Injection
- Propofol group (Active Comparator): 1. Background oxycodone injection: Slowly inject oxycodone(0.05mg/kg) intravenously. Three minutes (± 1min) after the end of oxycodone injection , begin sedation induction as follows.
  2. Sedation induction before EUS-FNA/FNB: the initial dose of propofol is 1.5-2.0 mg/kg, and the intravenous injection time is about 1 minute. If the subject's MOAA/S score is 1 point or below after the initial dose, EUS-FNA/FNB can be started; if the degree of sedation is insufficient, additional propofol(0.5 mg/kg each time) is allowed. The injection time of additional propofol is not less than 15 seconds, and the time interval between each additional administration is ≥ 2 minutes.
  3. Maintenance of sedation: In order to maintain the MOAA/S≤1, the investigator can decide to add propofol 0.5mg/kg each time, and the intravenous injection time should not be less than 15 seconds, with an additional administration interval of ≥ 2 minutes.
  Interventions: Drug: Propofol Injection

INTERVENTIONS:
Drug: Remimazolam Injection — The experimental group was sedated with remimazolam
  Arms: Remimazolam group
Drug: Propofol Injection — The control group was sedated with propofol
  Arms: Propofol group

SUMMARY:
This study aims to compare the safety and efficacy of remimazolam and propofol in EUS-FNA/FNB sedation. This study is a prospective, single-blind study. We plan to enroll 264 patients undergoing EUS-FNA and divide them into two groups. The experimental group was sedated with remimazolam, and the control group was sedated with propofol; safety and efficacy parameters such as intraoperative blood pressure, finger pulse oxygen, heart rate and sedation success rate would be compared. We hypothesized that patients in the experimental group would be superior in terms of safety parameters; the two would be equal in terms of sedation success.

DETAILED DESCRIPTION:
Endoscopic ultrasonography-guided fine needle aspiration/biopsy (EUS-FNA/FNB) is an important basis for the diagnosis of lesions in the upper gastrointestinal tract and adjacent organs, and plays an important role in the diagnosis of gastrointestinal tumors. Sedation is the key to a successful EUS-FNA/FNB procedure. However, intraoperative sedation in EUS-FNA/FNB is difficult and challenging. First, EUS-FNA/FNB requires a relatively long operation time and is prone to sedation-related adverse events, such as cardiovascular and cerebrovascular accidents. Second, EUS-FNA/FNB requires weakened gastrointestinal motility, thus deeper sedation is required during the operation; thirdly, the ultrasound probe used in EUS-FNA/FNB surgery is thicker than that of ordinary gastroscopes, which requires better cooperation from the patient. Therefore, the rational use of anesthesia drugs during surgery is required to ensure safety.

In current clinical studies, propofol is mostly used for anesthesia in patients undergoing EUS-FNA/FNB. In recent years, the defects of propofol for EUS sedation have gradually emerged, and its respiratory and circulatory inhibition effects have gradually caused researchers to worry. At present, propofol is still a commonly used EUS sedative drug, but with the improvement of people's requirements for sedation quality, its safety gradually cannot meet the demand. Therefore, it is the general trend to explore new EUS-FNA intraoperative sedation schemes.

Remimazolam is one of the new alternative drugs. Remimazolam is a new type of short-acting sedative-hypnotic drug, which has little inhibition on the respiratory system, less impact on hemodynamics, rapid onset of action, short half-life, rapid recovery, and no accumulation after long-term infusion. Thus, remimazolam is an effective drug for induction and maintenance of general anesthesia.

This study aims to compare the safety and efficacy of remimazolam and propofol in EUS-FNA/FNB sedation. This study is a prospective, single-blind interventional study. We plan to enroll 264 patients undergoing EUS-FNA and divide them into two groups. The experimental group was sedated with remimazolam, and the control group was sedated with propofol; safety and efficacy parameters such as intraoperative blood pressure, finger pulse oxygen, heart rate and sedation success rate would be compared. We hypothesized that patients in the experimental group would be superior in terms of safety parameters; the two would be equal in terms of sedation success.

This study is divided into the following steps:

1. Informed consent and participant recruitment First of all, inform the patients of the source, purpose, significance, and possible benefits and risks of participating in this study, so that patients can decide whether to participate after they have a full understanding. Patients who participated voluntarily signed the informed consent form. Eligible patients (n=264) would be selected according to the inclusion and exclusion criteria.
2. Information collection and participant screening Collect participant information, including name, gender, age, hospital number, enrollment date, education background, occupation, smoking status, drinking status, ASA classification, height, weight, lesion location, comorbidities (if any), medical history, physical examination results, laboratory examination results and imaging findings. Among them, physical examination results include general condition, upper limb skin, head, chest, abdomen, and necessary neurological examination results; laboratory results include blood routine, liver function, renal function, blood biochemistry, and coagulation routine. Imaging examinations are abdominal CT and other examination results that can reflect the location and size of the lesions.
3. Randomization With the help of the random number table pre-generated by SPSS20.0 software, participants would be divided into two groups (1:1). The sedation regimen is determined according to the random number obtained by the patient's lottery. The randomization process was completed by the designated study designer. Neither the patients nor the endoscopist knew the grouping status.
4. EUS-FNA/FNB information collection and preoperative preparation Collect operation information, including probe type, operation type, operator qualifications, operation indications, anesthesiologist qualifications, etc.

The patient fasted for at least 6 hours before the operation. Before the operation, the patient took 5ml of 2% lidocaine for topical anesthesia. Inhale oxygen for the patient (4L/min). The patient was placed in the left lateral decubitus position, connected to an ECG monitor, and venous access was established through the vein of the hand. The outpatient operating room is equipped with emergency facilities and equipment (emergency medicines, simple breathing balloons and masks, endotracheal intubation equipment and anesthesia machines).

5. Sedation induction and maintenance

1. Sedation protocol

   Remimazolam group:

   Background oxycodone injection: Slowly inject oxycodone(0.05mg/kg) intravenously. Three minutes (± 1min) after the end of oxycodone injection, begin sedation induction as follows.

   Sedation induction before EUS-FNA/FNB: the initial dose of remimazolam is 0.15-0.2 mg/kg, and the intravenous injection time is about 1 minute. If the subject's MOAA/S score is 1 point or below after the initial dose, EUS-FNA/FNB can be started; if the degree of sedation is insufficient, additional remimazolam(0.05 mg/kg each time) is allowed. The injection time of additional remimazolam is not less than 15 seconds, and the time interval between each additional administration is ≥ 2 minutes.

   Maintenance of sedation: In order to maintain the MOAA/S≤1, the investigator can decide to add remimazolam 0.05mg/kg each time, and the intravenous injection time should not be less than 15 seconds, with an additional administration interval of ≥ 2 minutes.

   Propofol group:

   Background oxycodone injection: Slowly inject oxycodone(0.05mg/kg) intravenously. Three minutes (± 1min) after the end of oxycodone injection , begin sedation induction as follows.

   Sedation induction before EUS-FNA/FNB: the initial dose of propofol is 1.5-2.0 mg/kg, and the intravenous injection time is about 1 minute. If the subject's MOAA/S score is 1 point or below after the initial dose, EUS-FNA/FNB can be started; if the degree of sedation is insufficient, additional propofol(0.5 mg/kg each time) is allowed. The injection time of additional propofol is not less than 15 seconds, and the time interval between each additional administration is ≥ 2 minutes.

   Maintenance of sedation: In order to maintain the MOAA/S≤1, the investigator can decide to add propofol 0.5mg/kg each time, and the intravenous injection time should not be less than 15 seconds, with an additional administration interval of ≥ 2 minutes
2. Judgment of sedation failure After the sedation inducement, if more than 5 additional doses are injected in any 15-minute time period, it is considered as a sedation failure. The anesthesiologist should use other sedative rescue measures (such as propofol, etc.) to maintain. After the additional bolus of the sedative, if the participant is still unable to cooperate due to physical movement or other reasons, but the interval between the next additional bolus does not reach 2 minutes, the anesthesiologist can decide to give the subject other sedative rescue measures (such as propofol, etc.) .In this case, failed sedation should be judged due to the use of sedative rescue measures.
3. Treatment protocol for adverse events The most likely adverse events in the study were respiratory depression, hypotension, and bradycardia. The corresponding treatment process is as follows: when the pulse oxygen saturation drops below 90% and does not recover spontaneously, the anesthesiologist will perform a 30-second chin lift operation; if blood oxygen saturation still cannot recover, increase the oxygen flow to 6L/min and the anesthesiologist compress the chest for assisted breathing; after 1 minute of observation, if there is still no recovery, a oxygen mask should be used; if it still cannot recover, perform mechanical ventilation or tracheal intubation. Hypotension was corrected with ephedrine (5 mg/time, intravenously) and bradycardia with atropine (0.5 mg/time, intravenously).

6. EUS-FNA/FNB operation and postoperative recovery EUS-FNA/FNB should perform according to routine procedures. After EUS-FNA/FNB procedure, patients were monitored in the postoperative recovery room until the modified Alderte score was 9 or greater before patients were allowed to leave. Patients will fill out the Modified Brice Questionnaire before departure.

7. Follow-up of patients 1-3 days after operation The patients were followed up 1-3 days after EUS/FNA-FNB to investigate the occurrence of adverse events and re-measure the changes of vital signs.

8. Data recording The patient's heart rate, systolic blood pressure, diastolic blood pressure, pulse oxygen saturation and MOAA/S score would be recorded every three minutes. Record the occurrence of adverse events, specific adverse event types, treatment methods and duration. 3) Record the total dosage of propofol or remimazolam after the operation.

ELIGIBILITY:
Inclusion Criteria:

1. Age: ≥18 years old and ≤75 years old
2. BMI: 18kg/m^2<BMI<30kg/m^2;
3. Body weight: 40kg<weight<120kg
4. Patients who intend and qualified to undergo sedated EUS-FNA/FNB.
5. Clearly understand, voluntarily participate in the research, and sign the informed consent form.

Exclusion Criteria:

1. Patients who are not suitable for sedated EUS-FNA/FNB for any reason (e.g. cardiovascular disease)
2. Patients have abnormal liver function, AST and/or ALT≥2.5×ULN, TBIL≥1.5×ULN;
3. Patients have abnormal renal function, urea or blood urea nitrogen≥1.5×ULN, serum creatinine≥1.0 ×ULN
4. Those who are allergic to benzodiazepines, opioids, propofol or lidocaine.
5. Patients have contraindications for benzodiazepines, opioids, propofol or lidocaine.
6. Patients have benzodiazepines, opioids, propofol, lidocaine suspected narcotic drug abuse history and pain drug or sedative abuse.
7. Patients have history of drug use and/or alcoholism within 2 years before the start of the period. Alcoholism means drinking more than 2 units of alcohol on average per day (1 unit = 360 mL of beer or 45 mL of liquor with an alcohol content of 40% or 150 mL of wine)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 264 (Estimated)
Dates: Start 2021-08-01 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Cardiopulmonary adverse event incidence | The whole EUS-FNA/FNB procedure
  The occurrence of any one of the following reactions was recorded as "Cardiopulmonary Adverse Event", and the cardiopulmonary adverse event incidence was defined as the proportion of the subjects with cardiopulmonary adverse events in each group. Cardiopulmonary adverse events were defined as: any of the following conditions occurred during the operation: 1. respiratory depression: oxygen saturation <90%, or breathing <8 times/min; 2. apnea: respiratory airflow stopped for more than 15s; 3. hypotension: systolic blood pressure decrease greater than 20% of baseline systolic blood pressure; 4. hypertension: systolic blood pressure increase greater than 20% of baseline systolic blood pressure; 5. tachycardia: heart rate>100bpm for 1 minute or more; 6. bradycardia: HR<50, lasting 1 minute or more

SECONDARY OUTCOMES:
Adverse event incidence | The whole EUS-FNA/FNB procedure
  The respective incidence of each adverse event that occurred during the EUS-FNA/FNB procedure, such as the incidence of cough or body movement.
Sedation success rate: | The whole EUS-FNA/FNB procedure
  Sedation success was defined as: completion of the entire procedure; no sedative rescue medication administered; ≤5 additional doses in any 15-minute period from the end of the initial dose of the trial drug. The sedation success rate was defined as the proportion of subjects in the group who were successfully sedated.

OTHER OUTCOMES:
Dosage of sedations | The whole EUS-FNA/FNB procedure
  The total dosage of remimazolam or propofol and the dosage per kilogram of body weight.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoyan Wang, Doctor, Principal Investigator — The Third Xiangya Hospital of Central South University
Locations (1):
- The Third Xiangya Hospital of Central South University, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: No
Some data underlying this trial cannot be shared publicly due to protection of participant's privacy.

REFERENCES:
- [Background] Behrens A, Kreuzmayr A, Manner H, Koop H, Lorenz A, Schaefer C, Plauth M, Jetschmann JU, von Tirpitz C, Ewald M, Sackmann M, Renner W, Kruger M, Schwab D, Hoffmann W, Engelke O, Pech O, Kullmann F, Pampuch S, Lenfers B, Weickert U, Schilling D, Boehm S, Beckebaum S, Cicinnati V, Erckenbrecht JF, Dumoulin FL, Benz C, Rabenstein T, Haltern G, Balsliemke M, de Mas C, Kleber G, Pehl C, Vogt C, Kiesslich R, Fischbach W, Koop I, Kuehne J, Breidert M, Sass NL, May A, Friedrich C, Veitt R, Porschen R, Ellrichmann M, Arlt A, Schmitt W, Dollhopf M, Schmidbaur W, Dignass A, Schmitz V, Labenz J, Kaiser G, Krannich A, Barteska N, Ell C. Acute sedation-associated complications in GI endoscopy (ProSed 2 Study): results from the prospective multicentre electronic registry of sedation-associated complications. Gut. 2019 Mar;68(3):445-452. doi: 10.1136/gutjnl-2015-311037. Epub 2018 Jan 3. PMID 29298872
- [Background] Pagano N, Arosio M, Romeo F, Rando G, Del Conte G, Carlino A, Strangio G, Vitetta E, Malesci A, Repici A. Balanced Propofol Sedation in Patients Undergoing EUS-FNA: A Pilot Study to Assess Feasibility and Safety. Diagn Ther Endosc. 2011;2011:542159. doi: 10.1155/2011/542159. Epub 2011 Jul 12. PMID 21785561
- [Background] Fatima H, DeWitt J, LeBlanc J, Sherman S, McGreevy K, Imperiale TF. Nurse-administered propofol sedation for upper endoscopic ultrasonography. Am J Gastroenterol. 2008 Jul;103(7):1649-56. doi: 10.1111/j.1572-0241.2008.01906.x. Epub 2008 Jun 28. PMID 18557709
- [Background] Nayar DS, Guthrie WG, Goodman A, Lee Y, Feuerman M, Scheinberg L, Gress FG. Comparison of propofol deep sedation versus moderate sedation during endosonography. Dig Dis Sci. 2010 Sep;55(9):2537-44. doi: 10.1007/s10620-010-1308-0. Epub 2010 Jul 16. PMID 20635148
- [Background] Kim MG, Park SW, Kim JH, Lee J, Kae SH, Jang HJ, Koh DH, Choi MH. Etomidate versus propofol sedation for complex upper endoscopic procedures: a prospective double-blinded randomized controlled trial. Gastrointest Endosc. 2017 Sep;86(3):452-461. doi: 10.1016/j.gie.2017.02.033. Epub 2017 Mar 8. PMID 28284883
- [Background] Heuss LT, Schnieper P, Drewe J, Pflimlin E, Beglinger C. Risk stratification and safe administration of propofol by registered nurses supervised by the gastroenterologist: a prospective observational study of more than 2000 cases. Gastrointest Endosc. 2003 May;57(6):664-71. doi: 10.1067/mge.2003.191. PMID 12709694
- [Background] Dewitt J, McGreevy K, Sherman S, Imperiale TF. Nurse-administered propofol sedation compared with midazolam and meperidine for EUS: a prospective, randomized trial. Gastrointest Endosc. 2008 Sep;68(3):499-509. doi: 10.1016/j.gie.2008.02.092. Epub 2008 Jun 17. PMID 18561925
- [Background] Trummel JM, Surgenor SD, Cravero JP, Gordon SR, Blike GT. Comparison of differing sedation practice for upper endoscopic ultrasound using expert observational analysis of the procedural sedation. J Patient Saf. 2009 Sep;5(3):153-9. doi: 10.1097/PTS.0b013e3181b53f80. PMID 19927048
- [Background] Amornyotin S, Leelakusolvong S, Chalayonnawin W, Kongphlay S. Age-dependent safety analysis of propofol-based deep sedation for ERCP and EUS procedures at an endoscopy training center in a developing country. Clin Exp Gastroenterol. 2012;5:123-8. doi: 10.2147/CEG.S31275. Epub 2012 Jul 9. PMID 22826640
- [Background] Yusoff IF, Raymond G, Sahai AV. Endoscopist administered propofol for upper-GI EUS is safe and effective: a prospective study in 500 patients. Gastrointest Endosc. 2004 Sep;60(3):356-60. doi: 10.1016/s0016-5107(04)01711-0. PMID 15332023
- [Background] Ye L, Xiao X, Zhu L. The Comparison of Etomidate and Propofol Anesthesia in Patients Undergoing Gastrointestinal Endoscopy: A Systematic Review and Meta-Analysis. Surg Laparosc Endosc Percutan Tech. 2017 Feb;27(1):1-7. doi: 10.1097/SLE.0000000000000373. PMID 28079763
- [Background] Wang F, Zhou Q, Shen M, Quan J, Chen J, Shi J, Zou X. Efficacy and safety of remimazolam in procedural sedation and analgesia: A protocol for systematic review and meta analysis. Medicine (Baltimore). 2020 Jul 2;99(27):e20765. doi: 10.1097/MD.0000000000020765. PMID 32629656
- [Background] Pastis NJ, Yarmus LB, Schippers F, Ostroff R, Chen A, Akulian J, Wahidi M, Shojaee S, Tanner NT, Callahan SP, Feldman G, Lorch DG Jr, Ndukwu I, Pritchett MA, Silvestri GA; PAION Investigators. Safety and Efficacy of Remimazolam Compared With Placebo and Midazolam for Moderate Sedation During Bronchoscopy. Chest. 2019 Jan;155(1):137-146. doi: 10.1016/j.chest.2018.09.015. Epub 2018 Oct 4. PMID 30292760
- [Background] Borkett KM, Riff DS, Schwartz HI, Winkle PJ, Pambianco DJ, Lees JP, Wilhelm-Ogunbiyi K. A Phase IIa, randomized, double-blind study of remimazolam (CNS 7056) versus midazolam for sedation in upper gastrointestinal endoscopy. Anesth Analg. 2015 Apr;120(4):771-80. doi: 10.1213/ANE.0000000000000548. PMID 25502841
- [Background] Pambianco DJ, Borkett KM, Riff DS, Winkle PJ, Schwartz HI, Melson TI, Wilhelm-Ogunbiyi K. A phase IIb study comparing the safety and efficacy of remimazolam and midazolam in patients undergoing colonoscopy. Gastrointest Endosc. 2016 May;83(5):984-92. doi: 10.1016/j.gie.2015.08.062. Epub 2015 Sep 9. PMID 26363333
- [Background] Rex DK, Bhandari R, Desta T, DeMicco MP, Schaeffer C, Etzkorn K, Barish CF, Pruitt R, Cash BD, Quirk D, Tiongco F, Sullivan S, Bernstein D. A phase III study evaluating the efficacy and safety of remimazolam (CNS 7056) compared with placebo and midazolam in patients undergoing colonoscopy. Gastrointest Endosc. 2018 Sep;88(3):427-437.e6. doi: 10.1016/j.gie.2018.04.2351. Epub 2018 Apr 30. PMID 29723512
- [Background] Uzman S, Gurbulak B, Gurbulak EK, Donmez T, Hut A, Yildirim D. A comparison of propofol and midazolam/meperidine sedation in upper gastrointestinal endoscopy. Wideochir Inne Tech Maloinwazyjne. 2016;11(3):178-185. doi: 10.5114/wiitm.2016.61521. Epub 2016 Jul 29. PMID 27829941
- [Background] Kashiwagi K, Hosoe N, Takahashi K, Nishino H, Miyachi H, Kudo SE, Martin JF, Ogata H. Prospective, randomized, placebo-controlled trial evaluating the efficacy and safety of propofol sedation by anesthesiologists and gastroenterologist-led teams using computer-assisted personalized sedation during upper and lower gastrointestinal endoscopy. Dig Endosc. 2016 Sep;28(6):657-64. doi: 10.1111/den.12678. Epub 2016 Jun 29. PMID 27176122

DOCUMENTS (3):
  • Study Protocol (2022-05-10): https://cdn.clinicaltrials.gov/large-docs/97/NCT05437497/Prot_000.pdf
  • Statistical Analysis Plan (2022-05-10): https://cdn.clinicaltrials.gov/large-docs/97/NCT05437497/SAP_001.pdf
  • Informed Consent Form (2022-05-10): https://cdn.clinicaltrials.gov/large-docs/97/NCT05437497/ICF_002.pdf